CLINICAL TRIAL: NCT06608680
Title: Timing and Facilitation Effects of Theta-Burst Stimulation in the Reading and Language Systems
Brief Title: Timing and Facilitation Effects of Theta-Burst Stimulation in the Reading and Language Networks
Acronym: TAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Rachael Marie Harrington, Assistant Professor, Georgia State University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: H23282
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Reading; Language; Control Subjects
Keywords: transcranial magnetic stimulation; TMS; MRI; Reading; Language
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTBS/Sham (Experimental): Adults age 18-30 with typical reading and language abilities
  Interventions: Behavioral: iTBS; Behavioral: Sham Stimulation
- cTBS/Sham (Experimental): Adults age 18-30 with typical reading and language abilities
  Interventions: Behavioral: cTBS; Behavioral: Sham Stimulation

INTERVENTIONS:
Behavioral: iTBS — Excitatory stimulation of supramarginal gyrus
  Arms: iTBS/Sham
Behavioral: cTBS — Inhibitory stimulation to supramarginal gyrus
  Arms: cTBS/Sham
Behavioral: Sham Stimulation — Sham stimulation of supramarginal gyrus

SUMMARY:
The purpose of this study is to understand how transcranial magnetic stimulation affects how quickly, easily, and accurately a person read. Transcranial magnetic stimulation is a technique that uses magnetic fields to briefly affect how well certain brain regions function. The investigators would like to better understand how long the effects of transcranial magnetic stimulation occur in the reading system and at what point the effect is strongest in this system. The main questions it aims to answer are:

1. At what point after stimulation are the greatest effects on behavior seen
2. How excitatory and inhibitory stimulation affect behavior

Researchers will compare stimulation types against a sham condition to see effects on reading and language behavior.

Participants will be asked to

* undergo reading, language, and cognitive testing
* receive an MRI
* receive TMS stimulation
* perform language, reading, and motor tasks

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a minimum of low average intellectual functioning (>=80) on at least one subscale on the Wechsler Abbreviated Scale of Intelligence-2 (WASI-2; Wechsler, 2011) to be included.
* Within a normal range of reading skills as >85 on the Test of Word Reading Efficiency - Second Edition (TOWRE-2; Torgesen et al., 2012) and the Woodcock-Johnson IV Tests of Achievement (WJ-IV; Schrank et al., 2014)
* Individuals with a documented history of learning disability will not be included. This will be determined via demographics questionnaire.
* Subjects must be between the ages of 18 and 30 to be included. This will be determined via demographics questionnaire.
* Because reading is critically linked to language, only individuals who are native speakers of English will be included in the study. This will be determined via demographics questionnaire.
* The reading network is typically localized to the left side of the brain. However, left-handed individuals may have different brain lateralization, introducing an important confound to the study. Therefore, only right-handed individuals will be included in the study. This will be determined via demographics questionnaire.
* Individuals who have hearing deficits (>25dB at 500+ Hz), visual deficits (>20/40), serious emotional problems, certain neurological conditions (e.g., uncontrolled seizure disorders) will not be included. This will be determined via CABI Screening Forms and Demographics Questionnaire.
* Individuals with certain metals in their bodies or with certain health conditions will not be included. If an individual has braces on their teeth, a cardiac pacemaker; hearing aid; other metal in their body or eyes (which may include certain metallic-embedded tattoos), including but not limited to pins, screws, shrapnel, plates, dentures or other metal objects they will not be included. This will be determined via CABI Screening forms.
* Individuals with MRI Screening and Contraindication Forms which do not pass MRI Tech review will not be included.
* Individuals with TMS Screening Forms which do not pass TMS Tech review will not be included.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Phonological Decoding Reaction Time | Four time points after each stimulation (20, 40, 60 and 80 minutes after stimulation)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared via the COINS platform